CLINICAL TRIAL: NCT00794963
Title: Aggressive Treatment of Metabolic Syndrome in Patients Treated With Clozapine for Schizophrenia
Brief Title: Aggressive Treatment of Metabolic Syndrome in Patients Receiving Clozapine for Schizophrenia
Acronym: ATOMICS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Peter Manu, Professor of Medicine and Psychiatry, Hofstra NS-LIJ School of Medicine, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-177
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Results first posted 2011-11-18 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2011-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Pravastatin; Fenofibrate; Metformin; Orlistat; Irbesartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated care (Experimental): Provide on-site internal medicine evaluation, treatment and follow up of metabolic syndrome for patients in Clozapine Clinic
  Interventions: Drug: Pravastatin, Fenofibrate, Metformin, Orlistat, irbesartan
- Usual Care (Other): Follow the 8-month outcome of schizophrenia patients with metabolic syndrome treated in the community
  Interventions: Other: As selected by community physician

INTERVENTIONS:
Drug: Pravastatin, Fenofibrate, Metformin, Orlistat, irbesartan — The intervention in the 4 patients consisted in dietary recommendations, advice regarding increasing physical activity, and use of Orlistat 60 mg three times daily. No other drugs were prescribed.
  Arms: Integrated care
Other: As selected by community physician — As selected by community physician
  Arms: Usual Care

SUMMARY:
Schizophrenia patients treated with clozapine have a high prevalence of obesity-related metabolic syndrome. The condition is often poorly treated and may lead to the emergence of coronary heart disease and type 2 diabetes. The study will investigate whether structured treatment provided at the site of the outpatient psychiatric clinic of metabolic syndrome in this population will decrease the severity of metabolic syndrome as compared with usual care received by these patients in the community.

DETAILED DESCRIPTION:
Background

Compared with the general population, patients with schizophrenia have an increased risk of death from atherosclerotic cardiovascular diseases (ASCVD) that reflect coronary heart disease, stroke and peripheral vascular disease (Newcomer, 2007). Among the factors contributing to the increased prevalence of ASCVD in schizophrenia are a) unhealthy lifestyle (cigarette smoking, lack of physical activity, increased consumption of calorie-dense foods rich in saturated fats and carbohydrates), b) genetic vulnerability to glucose intolerance and diabetes; c) metabolic side-effects of psychotropic drugs; and d) lack of access or compliance with community-based medical care, particularly clozapine or olanzapine. Biologically, the common pathway leading to increased risk of ASCVD in schizophrenia is the metabolic syndrome, an entity defined as 3 or more of the following 5 characteristics: abdominal obesity, increased blood pressure, increased fasting glucose, increased levels of triglycerides and abnormally low levels of high-density lipoprotein cholesterol. The prevalence of metabolic syndrome in schizophrenia ranges form 29% to 63% and is significantly greater than the frequency of 21% in the general population (Correll et al., 2006). As in the general population, the metabolic syndrome of patients with schizophrenia is explained by increased intraabdominal adiposity leading to insulin resistance and excess of circulating free fatty acids which are converted into triglyceride-rich lipoproteins with atherogenic potential.

The treatment of metabolic syndrome relies primarily on therapeutic lifestyle changes aiming to reduce weight, decrease intake of saturated fats and carbohydrates with high glycemic index, eliminate smoking, and increase physical activity. Drug therapy is required for the patients who fail to respond to lifestyle changes and the American Heart Association (AHA) has published detailed guidelines for the pharmacologic management of metabolic syndrome (Grundy et al., 2005). These guidelines are based on research indicating substantial improvement in the risk of ASCVD of patients with metabolic syndrome treated with metformin and acarbose for impaired glucose tolerance; statins, fibrates and nicotinic acid for lipid abnormalities; angiotensin receptor blockers for increased blood pressure; and sibutramine and orlistat for weight management. Some of these interventions (e.g., metformin and sibutramine for weight management) have been completed in research settings with small samples of patients with schizophrenia (Henderson et al., 2005; Wu et al., 2008) and have produced promising results. However, treatment trials using the comprehensive AHA guidelines have not yet been conducted in schizophrenics with metabolic syndrome.

Current Standard of Care at Zucker Hillside Hospital

The Aftercare Clinic at Zucker Hillside Hospital has the oldest Clozapine Clinic in the U.S. Opened in 1987, the Clozapine Clinic has a current enrollment of 230 adult patients. According to hospital policy, all Clozapine Clinic patients must have an annual physical evaluation and laboratory tests for the detection of obesity, dyslipidemia, glucose intolerance, hypertension and metabolic syndrome. The mandatory physical examinations are performed by each patient's outside physician or by the Clinic's Nurse Practitioners. Laboratory testing is performed at Long Island Jewish Medical Center's laboratories. The physical examinations and laboratory findings are reviewed by each patient's psychiatrists. Patients with physical or laboratory abnormalities are referred for care to internal medicine specialists (i.e., general internal medicine, endocrinology, cardiology) in private practice or to the appropriate outpatient clinics at Long Island Jewish Medical Center as deemed necessary by their psychiatrists. At the present time, it is not known how many schizophrenia patients with metabolic syndrome treated in the Aftercare Program (outpatient clinic) at ZHH receive care according to the standard defined by the American Heart Association.

Objective

We plan to evaluate the effect of application of AHA guidelines for the treatment of metabolic syndrome in patients with schizophrenia who are receiving clozapine, an antipsychotic known to produce weight gain and metabolic abnormalities in a majority of patients (Newcomer, 2006). The study will include only outpatients receiving care in the Clozapine Clinic. .

The study's primary aim is to compare the effectiveness of managing metabolic syndrome in schizophrenia at the site of psychiatric outpatient services (integrated care) with treatment obtained and coordinated by the patients Hillside psychiatrist (usual care). We propose that Integrated care will remove access barriers, improve compliance, enhance communication between psychiatry and internal medicine providers, and facilitate education for weight management and smoking cessation. The management of metabolic syndrome for patients receiving integrated care will adhere to the AHA guidelines (Grundy et al., 2005) which describe dietary, exercise and pharmacologic interventions that have been extensively validated in the general population. All of the medications suggested in the guidelines have been FDA-approved for the individual components of metabolic syndrome. The 'usual care' group will receive the current standard of care set by Hillside Hospital.

Importance of the Study

This is the first randomized trial of a "no-barriers" model of medical care for an underserved and vulnerable mentally ill population. To increase homogeneity of the study population and significance of the expected difference between integrated and usual care, the study will assess only patients with the same psychiatric diagnosis (schizophrenia), treated with the same psychotropic (clozapine) in a single, well-established outpatient setting. The duration of the study is adequate to demonstrate whether the metabolic syndrome components respond to life style modification and /or specific pharmacological intervention.

Research Design and Methods

Hypothesis

Integrated, on-site, medical management of metabolic syndrome in patients with schizophrenia is superior to usual care in the community, primarily because it will remove barriers related to access to medical providers and increase compliance with drug therapy and laboratory testing. The improvement will lead to decreased frequency of metabolic syndrome in the sample, decreased risk of future ASCVD events (as predicted by AHA-recommended instruments), decreased waist circumference, fasting glucose, blood pressure and triglyceride levels and increased levels of HDL.

ELIGIBILITY:
Inclusion Criteria:

* patients with schizophrenia treated with clozapine; age 19-79

Exclusion Criteria:

* pregnant women, personal history of/or comorbid eating disorders

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Zucker Hillside Hospital, Glen Oaks, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Integrated Care | Usual Care
Started | 4 | 4
Completed | 3 | 0
Not Completed | 1 | 4
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrated Care | Usual Care | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (4.8) | 43.5 (5.6) | 48.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Time Frame: baseline and 8 months
Population: 4 participants in usual care arm did not return for follow-up and were not available for analysis; 1 participant in the integrated care group was lost to follow-up
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Integrated Care | Usual Care
Number analyzed (Participants) | 3 | 0
pounds | 11 (5.6) |

ADVERSE EVENTS:
Arm/Group | Integrated Care | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No